CLINICAL TRIAL: NCT06153784
Title: Long-Term Assessment of Thalidomide and Hydroxyurea Combination Therapy in β-Thalassemia Patients
Brief Title: Thalidomide and Hydroxyurea Combination in β-Thalassemia Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Karachi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-0428
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Thalassemia, Beta
MeSH Terms: conditions — beta-Thalassemia | interventions — Hydroxyurea; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of hydroxyurea and thalidomide (Experimental): Hydroxyurea was continued at a dose of 10-20 mg/kg/day for 6 months and then thalidomide was added orally at a dose of 2-5mg/kg/day.
  Interventions: Drug: Hydroxyurea and Thalidomide

INTERVENTIONS:
Drug: Hydroxyurea and Thalidomide — Evaluation of hydroxyurea and thalidomide combination use in beta-thalassemia patients

SUMMARY:
Objectives

Primary objective:

• To determine the efficacy and safety of the combination therapy of Hydroxyurea and thalidomide in beta-thalassemia patients.

Secondary objective:

• To determine the change in liver and spleen size of beta-thalassemia patients on the combination therapy.

A single-arm non-randomized trial to evaluate the efficacy and safety of combination therapy of hydroxyurea and thalidomide in beta-thalassemia patients. Participants were monitored for six months on Hydroxyurea alone and then the combination therapy of hydroxyurea and thalidomide was started. Findings of physical examination, vital signs, laboratory, and ultrasound findings were recorded at baseline, during, and end of the study.

The assessment of treatment outcomes was conducted at the 1-year, 2-year, and 3-year follow-up points during the combination therapy period, categorizing patients as either "good responders," "responders," or "non-responders."

DETAILED DESCRIPTION:
This study is conducted to evaluate the long-term efficacy and safety of the combination therapy of hydroxyurea and thalidomide in beta-thalassemia patients.

Monotherapy of Hydroxyurea was sustained at a daily dosage ranging from 10-20 mg/kg for a duration of 6 months, during which the treatment response was documented. After this initial 6-month period, thalidomide was introduced into the treatment regimen. Thalidomide was administered orally at bedtime, with an initial dosage of 2-5 mg/kg. An incremental dosing approach was employed for thalidomide, with individuals who exhibited an insufficient response to lower doses having their dosage increased to a maximum of 5 mg/kg. Additionally, aspirin was prescribed at a daily dosage of 2-4 mg/kg to mitigate the risk of thrombosis.

Blood transfusions were administered under specific conditions throughout the study. Transfusions were initiated if the Hb levels dropped below 7 g/dL or if patients exhibited symptoms or instability, regardless of their Hb levels. Patients who were undergoing iron chelation therapy (utilizing deferasirox, deferiprone, and/or deferoxamine) while on HU monotherapy continued this regimen throughout the combination therapy phase.

Throughout combination therapy, various assessments were conducted and documented, including blood transfusion events and comprehensive blood count evaluations, carried out at baseline, as well as during the 1-year, 2-year, and 3-year follow-up periods. Concurrently, safety parameters, such as urea and creatinine levels, liver function tests, and measurements of liver and spleen size, were consistently monitored and recorded.

Outcome:

Good responders were characterized as individuals who were previously reliant on blood transfusions while on hydroxyurea therapy but became transfusion-independent after the initiation of hydroxyurea and thalidomide combination therapy. Furthermore, patients who were already free from transfusions while on hydroxyurea therapy and demonstrated an increase in Hb levels exceeding 1 g/dL upon combination therapy were also classified as good responders.

Responders were defined as patients who, while receiving blood transfusions during hydroxyurea therapy, exhibited a substantial reduction of at least 50% in the volume of PRC transfusions over a span of 6 months after the onset of combination therapy.

Non-responders encompassed patients who were not reliant on transfusions during hydroxyurea therapy but did not display any significant enhancement in Hb levels following the commencement of combination therapy. Additionally, individuals who were dependent on transfusions but experienced less than a 50% reduction in PRC transfusion volume despite hydroxyurea and thalidomide combination therapy were also categorized as non-responders.

Safety:

The safety of the drug was evaluated based on the following parameters and the intervention was discontinued or put on hold if:

* Creatinine >1.1mg/dl, Urea >43mg/dl),
* Liver function (SGPT >35mg/L)
* Absolute Neutrophil counts<2*109/L
* Platelets < 100*109/L

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical and genetic diagnoses of β-thalassemia major and intermedia
2. Patients who showed partial response or a decline in response to hydroxyurea
3. Patients who are not candidates for the bone marrow transplant procedure

Exclusion Criteria:

1. Married Patients
2. Patients with comorbidities such as liver, cerebrovascular, cardiovascular, or kidney diseases
3. Patients allergic to the drug ingredients
4. Patients with mental disorders
5. Patients who are enrolled in other clinical trials
6. Patients with a history of venous or arterial thrombosis

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 603 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Response at different time intervals | 1-3 years on combination therapy
  Frequency of good responder, responder, and non-responder.
Change in laboratory levels | 1-3 years on combination therapy
  Mean changes in hemoglobin, platelets, leukocytes, urea, creatinine, and ferritin level from baseline
Change in the liver and spleen size | 1-3 years on combination therapy
  Mean changes in the liver and spleen size from baseline

SECONDARY OUTCOMES:
XmnI polymorphism | 1-3 years on combination therapy
  Comparison of XmnI polymorphism with outcome among patients who completed 1-year, 2-years, and 3-years of combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Saqib H Ansari, Phd, Principal Investigator — Children's Hospital Karachi Sindh, Pakistan
Locations (1):
- Children's Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No